CLINICAL TRIAL: NCT06027567
Title: Glucagon-like Peptide-1 Receptor (GLP-1R) Analogue Assisted Rapid Weight Loss Program As Treatment of Idiopathic Intracranial Hypertension
Brief Title: The Effect of an Anti-obesity Drug, Semaglutide, As Treatment in New-onset Idiopathic Intracranial Hypertension (IIH) Compared to Standard Weight Management (dietician) with Regards to Change in Weight and Intracranial Pressure
Acronym: IIH:DUAL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rigmor Højland Jensen (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Rigmor Højland Jensen, Professor in Neurology, Danish Headache Center
Organization: Danish Headache Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIH:DUAL
Record Dates: First submitted 2023-02-23; First posted 2023-09-07 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Intracranial Hypertension; Intracranial Pressure; Obesity; Pseudotumor Cerebri Syndrome; Papilledema; Weight Loss
Keywords: Idiopathic Intracranial Hypertension; Papilledema; Weight loss; Obesity; Pseudotumor Cerebri Syndrome; Intracranial Pressure
MeSH Terms: conditions — Pseudotumor Cerebri; Obesity; Papilledema; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Open label randomized controlled clinical treatment trial Patients are randomly assigned 1:1 to standard-of-care or intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): Semaglutide up-titration to 2.4 mg for 10 months initially combined with a Very Low Calorie Diet (800 kcal/day) for 8 weeks.
  Counselling by dietician Standard medical treatment of intracranial hypertension
  Interventions: Drug: Semaglutide; Dietary Supplement: Very Low Calorie Diet; Behavioral: Dietician counselling
- Standard care (dietician) (Active Comparator): Standard weight loss intervention Counselling by dietician Standard medical treatment of intracranial hypertension
  Interventions: Behavioral: Dietician counselling

INTERVENTIONS:
Drug: Semaglutide — Subcutaneous once-weekly injections of Semaglutide uptitrating to a maximum of 2.4 mg
  Other Names: Ozempic, Wegovy
  Arms: Semaglutide
Dietary Supplement: Very Low Calorie Diet — Very Low Calorie Diet (max 800 kcal/day) using Nupo Diet meal replacement products
  Arms: Semaglutide
Behavioral: Dietician counselling — Counselling by a dietician on weight loss through behavioural changes and life style intervention

SUMMARY:
50 patients with verified new-onset Idiopathic Intracranial Hypertension are randomly allocated to standard weight management (dietician counselling) or trial intervention consisting of subcutaneous injections with Semaglutide for 10 months combined, in the initial 8 weeks following diagnosis, with a Very Low Calorie-Diet (max 800 kcal/day)

DETAILED DESCRIPTION:
Idiopathic Intracranial Hypertension is primarily observed in obese female and weight management promotes disease control by yet unsettled mechanisms. Effective, fast and lasting weight loss is crucial, however, hard to achieve. Current weight management strategy in IIH in Denmark is counselling by a dietician. This study investigates whether an initial Very Low Calorie Diet (max 800 kcal/day) for 8 weeks following the diagnosis combined with GLP1-RA treatment throughout 10 months is tolerated and more efficient in achieving substantial weight loss and reduction of intracranial pressure. Furthermore, a number of secondary outcomes are measured including headache burden, quality of life, structure and function of the optic nerve, non-invasive surrogate markers of intracranial pressure, body fat mass, bone health, fatty liver disease and a range of cerebrospinal-, blood- and urine markers of i.a. the hormonal, inflammatory, metabolic, and headache biomarker profile.

The intervention may candidate as a future first-line treatment regime.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new onset definite IIH with papilledema and lumbar opening pressure ≥25 cm cerebrospinal fluid according to Friedmann diagnostic criteria
* BMI ≥ 27
* Use of contraceptive methods with failure rates of less than 1 % throughout the study period for group A and for at least an additional 2 months after cessation of Semaglutide
* Written, informed consent

Exclusion Criteria:

* Unable to provide written informed consent or participate
* Malignant IIH with visual threat that requires surgical intervention, i.e., cerebrospinal fluid diversion (shunting), optic nerve sheet fenestration or cerebral venous sinus stenting
* Pregnancy or breastfeeding
* Treatment with antidiabetics, blood-thinners or medication that may increase the risk of adverse events
* Diabetes, congestive heart failure, severe vascular disease, pancreatitis, severe ophthalmological disorders other than IIH (e.g. retinopathy)
* History or family history of thyroid carcinomas or Multiple Endocrine Neoplasias (MEN1/MEN2)
* History of bariatric surgery
* Known hypersensitivity to any contents of Semaglutide®
* Other severe/uncontrolled mental or physical disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Weight | 8 weeks
  Weight change (%)
Intracranial pressure | 8 weeks
  Change in lumbar opening pressure in cm cerebrospinal fluid measured by manometry
Intracranial pressure | 8 weeks
  Change in lumbar opening pressure (%)

SECONDARY OUTCOMES:
Weight | 10 months
  Weight change (%)
Intracranial Pressure | 10 months
  Change in lumbar opening pressure in cm cerebrospinal fluid measured by manometry
Intracranial Pressure | 10 months
  Change in lumbar opening pressure (%)
Quality of Life | 8 weeks + 10 months
  Change in total score of Quality of Life (psychological, social, physical, environmental) assessed by the World Health Organization Quality of Life Brief Version Questionnaire (0-100; 0 worst, 100 best)
Headache burden measured by HURT questionnaire | 8 weeks + 10 months
  Change in summation of scores in the questionnaire "Headache Under Response to Treatment Questionnaire" (HURT); 0-24 points were higher numbers are worse outcome
Change in Papilledema | 8 weeks + 10 months
  Change in Frisén Grade (0-5, 0 minimal, 5 worst)
Visual fields | 8 weeks + 10 months
  Perimetric mean deviation (decibel) by Humphrey automated perimetry
EDI-OCT | 8 weeks + 10 months
  Change in Papillary thickness (um) measured by Enhanced Depth Imaging Optical Coherence Tomography (EDI-OCT)
Optic disc elevation | Baseline + 8 weeks + 10 months
  Optic disc elevation (mm) measured by transorbital ultrasonography, (average of 3 scans of each eye with papilledema)
Remission | 8 weeks + 10 months
  Proportion of patients with abscence of papilledema with or without intracranial pressure <25 cm cerebrospinal fluid
Change in fat mass | 8 weeks + 10 months
  Change in body fat percentage measured by Dual Energy X-ray Absorptiometry compared to baseline
Total fat mass | Baseline + 8 weeks + 10 months
  Body fat percentage measured by Dual Energy X-ray Absorptiometry
Feasibility | 8 weeks + 10 months
  Drop-out rate (proportion of patients withdrawing from participation)
Need of intracranial pressure-lowering medication_1 | 8 weeks + 10 months
  Dose (mg) of intracranial pressure-lowering medication needed (Acetazolamide, Topiramate, diuretics)
Fatty liver prevalence | Baseline + 8 weeks + 10 months
  Prevalence of non-alcoholic fatty liver disease evaluated by ultrasonography (subjectively assessed density of liver parenchyma compared to hepatic perivascular density and renal density), assessed by an experienced radiologist with specialization in ultrasonography
Monthly headache days | Baseline + 8 weeks + 10 months
  Number of days with headache for the past 30 days preceding visit
Headche severity | Baseline + 8 weeks + 10 months
  Number of days with mild, moderate, and severy headache, respectively, in the past 30 days preceding visit
Headache medication - Acute analgesic use | Baseline + 8 weeks + 10 months
  Number of days with need of acute analgesic treatment for headache
Headache medication - preventive medication | Baseline + 8 weeks + 10 months
  Need of preventive medical treatment for headache
Optic nerve sheath diameter | Baseline + 8 weeks + 10 months
  Optic nerve sheath diameter (mm) measured by transorbital ultrasonography (average of 3 scans of each eye with papilledema)
Peripapillary capillary density | Baseline + 8 weeks + 10 months
  Change in peripapillary capillary density (ratio of pixels of perpapillary vessels and pixels in the foveal area evaluated by Optic Coherence Tomography Angiography
Peripapillary artery-to-venule ratio | Baseline + 8 weeks + 10 months
  Change in peripapillary artery-to-venule diameter ratio measured by confocal Scanning Laser Ophtalmoscopy
Truncal fat | Baseline + 8 weeks + 10 months
  Change in percentage of truncal adiposity measured by Dual Energy X-ray Absorptiometry
Android-gynoid-ratio | Baseline + 8 weeks and 10 months
  Change in ratio of Android versus gynoid fat percentage using Dual Energy X-ray Absorptiometry
Adverse events | 8 weeks + 10 months
  Number of adverse events overall, and sub-categorized into adverse events (AE) (any event happening during attachment to the project) and severe adverse events (SAE) in case of the following conditions: Hospitalization or prolongation of hospitalization, death, life-threatening or significant disability/incapacity
Need of intracranial pressure-lowering medication_2 | Baseline + 8 weeks + 10 months
  Number of patients in need of any intracranial pressure-lowering drug (Acetazolamide, Topiramate, diuretics)
Insulin like-Growth-Factor-1 | Baseline
  Level of Insulin like-Growth-Factor-1 in serum (ug/L) in women not taking estrogen-containing contraceptives.
Insulinlike Growth Factor Binding Protein-3 | Baseline
  Level of Insulinlike Growth Factor Binding Protein-3 in serum (ug/L) in women not taking estrogen-containing contraceptives.
Growth hormone | Baseline
  Level of growth hormone in serum ug(L) in women not taking estrogen-containing contraceptives.
Lutropin | Baseline
  Level of Lutropin in serum (IU/L) in women not taking estrogen-containing contraceptives.
Follitropin | Baseline
  Level of Follitropin in serum (IU/L) in women not taking estrogen-containing contraceptives.
Testosteron | Baseline
  Level of testosteron in serum (nmol/L) in women not taking estrogen-containing contraceptives.
Estradiol | Baseline
  Level of estradiol in serum (nmol/L) in women not taking estrogen-containing contraceptives.
Sex-Hormone Binding Globulin | Baseline
  Level of Sex-Hormone Binding Globulin in serum (nmol/L) in women not taking estrogen-containing contraceptives.
Anti-Müllerian Hormone | Baseline
  Level of Anti-Müllerian Hormone (pmol/L) in serum in women not taking estrogen-containing contraceptives.
Dehydroepiandrosterone | Baseline
  Level of Dehydroepiandrosterone (DHEAS) in serum (umol/L) in women not taking estrogen-containing contraceptives.
Androstenedion | Baseline
  Level of androstenedion (nmol/L) in serum in women not taking estrogen-containing contraceptives.
17-hydroxyprogesterone (mg/d) | Baseline
  Level of 17-hydroxyprogesterone (mg/d) in serum in women not taking estrogen-containing contraceptives.
Cortisol 0 min | Baseline
  Level of cortisol (nmol/L) in serum in women not taking estrogen-containing contraceptives.
Cortisol 30 min | Baseline
  Level of cortisol (nmol/L) in serum 30 minutes after stimulation with 0,25 mg SynACHTen in women not taking estrogen-containing contraceptives.
Pituitary adenylate cyclase-activating peptide (PACAP) Pituitary adenylate cyclase-activating peptide Pituitary adenylate cyclase-activating peptide | Baseline + 8 weeks + 10 months
  Level (picograms per milliliter in plasma and cerebrospinal fluid) of Pituitary adenylate cyclase-activating peptide (PACAP)
Calcitonin Gene Related Peptide | Baseline + 8 weeks + 10 months
  Calcitonin Gene Related Peptide (CGRP) level pg/mL (picograms per milliliter in plasma and cerebrospinal fluid)
Change in bone marker (CTX) | Baseline + 8 weeks + 10 months
  Change in carboxy-terminal collagen crosslinks (CTX) level (nanograms per liter)
Change in bone marker (PiNP) | baseline + 8 weeks + 10 months
  Change in procollagen type I N-propeptide (PiNP) level (micrograms per liter) compared to baseline
Regional bone density | Baseline + 8 weeks + 10 months
  Change in regional bone density in grams/square cm (g/cm2) and T- and Z-scores of hip and spine measured by Dual Energy X-ray Absorptiometry compared to baseline
Androgen metabolism_1 | Baseline + 8 weeks + 10 months
  Ratio between Etiocholanolone and Androsterone (ng/mg) in 24-hour urine
Androgen metabolism_2 | Baseline + 8 weeks + 10 months
  Ratio between 5-alpha-tetrahydrocortisol (5a-THF) and tetrahydrocortisol (THF) in 24-hour urine
Androgen metabolism_3 | Baseline + 8 weeks + 10 months
  Level of testosterone in 24-hour urine (ng/L)
Androgen metabolism_4 | Baseline + 8 weeks + 10 months
  Level of 3-alpha-androstanediol in 24-hour urine (nmol/L)
Androgen metabolism_5 | Baseline + 8 weeks + 10 months
  Level of 11-oxygenated androgens (11-OHA4) (pg/L) in 24-hour urine
Intrathecal Semaglutide | 10 months
  Level of semaglutide in cerebrospinal fluid (picomol/L)
Ammoniaemia_1 | Baseline + 8 weeks + 10 months
  Levels of plasma ammonium (umol/L)
Ammoniaemia_2 | Baseline + 8 weeks + 10 months
  Correlation between plasma ammonium (umol/L) and presence of fatty liver disease as indicated by liver ultrasonography
Ketosis | 8 weeks + 10 months
  Proportion of patients in ketosis measured by urine stix
Change in metabolic parameters | 8 weeks + 10 months
  Change in Homeostatic Model for Insulin Resistance (HOMA2IR) compared to baseline
Change in metabolic parameters | 8 weeks + 10 months
  Change in glycated hemoglobin (mmol/mol) compared to baseline

OTHER OUTCOMES:
Omics | Baseline + 8 weeks + 10 months
  Metabolomic and proteomic profile, exploratory analyses

CONTACTS AND LOCATIONS:
Overall Officials: Rigmor H Jensen, Professor, Study Director — Danish Headache Center
Locations (2):
- Denmark (2):
  - Headache clinic, Department of Neurology, Odense University Hospital, Odense, Odense
  - Danish Headache Center, Department of Neurology, Rigshospitalet, Glostrup Municipality

IPD SHARING:
Plan to Share IPD: No